CLINICAL TRIAL: NCT06314490
Title: Personalized Antisense Oligonucleotide Therapy for Rare Pediatric Genetic Disease: SCN2A
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); n-Lorem Foundation (Other)
Responsible Party: Principal Investigator, Olivia Kim-McManus, Professor, Neurosciences, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASOSCN2A
Record Dates: First submitted 2024-03-01; First posted 2024-03-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label (Experimental)
  Interventions: Drug: nL-SCN2A-002

INTERVENTIONS:
Drug: nL-SCN2A-002 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single pediatric participant with SCN2A associated developmental epileptic encephalopathy

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single pediatric participant with a de novo pathogenic gain of function SCN2A mutation associated with severe developmental epileptic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant's parent(s)/guardian(s)
* Ability to travel to the study site, adhere to study-related follow-up examinations and/or procedures, and provide access to participant's medical records.
* Genetically confirmed mutation

Exclusion Criteria:

• Use of an investigational medication within less than 5 half-lives of the drug at enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | Baseline to 24 months
  As measured by caregiver provided seizure diary
Motor function as measured by Dyskinetic Cerebral Palsy Functional Impact Scale | Baseline to 24 months
  The Dyskinetic Cerebral Palsy Functional Impact Scale (D-FIS) is an 18 item caregiver questionnaire that evaluates the impact of dyskinesia on daily functions. It is a validated assessment tool for children aged 2 years and 6 months to 18 years. It uses a 5-point ordinal scale, from 0 (no impact) to 4 (extreme impact), for each item and derives a total score from summing all 18 items. A higher score indicates more severe impact of dyskinesia and worse motor functioning.
Motor function as measured by the motor skills domain of Vineland Adaptive Behavior Scales | Baseline to 24 months
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3), is a standardized, validated, and reliable assessment tool designed to measure the adaptive behavior of individuals from birth through adulthood. The Vineland-3 Motor Skills domain evaluates gross and fine motor abilities in individuals from birth to age 9, offering insights into coordination, balance, mobility, and dexterity. The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better adaptive functioning.
Motor function as measured by the motor skills domain of Bayley Scales of Infant and Toddler Development | Baseline to 24 months
  The Bayley Scales of Infant and Toddler Development is a standardized, validated, and reliable assessment tool for evaluating developmental functioning in infants and toddlers. Its Motor Skills domain evaluates gross and fine motor abilities, including coordination, balance, and movement. The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better motor development.
Gastrointestinal assessment as measured by the Bristol Stool Chart | Baseline to 24 months
  The Bristol Stool Chart categorizes human feces into seven types, from Type 1 (severe constipation) to Type 7 (diarrhea), with Types 3 and 4 considered normal.

SECONDARY OUTCOMES:
Neurodevelopmental Function as measured by Aberrant Behavior Checklist | Baseline to 24 months
  The Aberrant Behavior Checklist (ABC) is an empirically developed scale tailored to measure psychiatric symptoms and behavioral disturbances in individuals with Intellectual and Developmental Disabilities (IDD). It contains five domains: Irritability, Agitation, & Crying; Lethargy/Social Withdrawal; Stereotypic Behavior; Hyperactivity/Noncompliance; and Inappropriate Speech. Each question is scored on a 4-point scale (0 = not a problem to 3 = severe problem) to assess severity. Total scores per subscale reflect the extent of behavioral challenges, with higher scores indicating greater severity.
Neurodevelopmental Function as measured by Observer-Reported Communication Ability Measure | Baseline to 24 months
  The Observer-Reported Communication Ability (ORCA) Measure is a questionnaire assessing communication abilities in individuals with neurodevelopmental disorders, significantly impacting verbal speech. It includes 84 questions, with 70 behavioral items across 22 concepts/functions and 14 descriptive items about individual communication methods, covering expressive, receptive, and pragmatic communication areas. The ORCA is validated for Angelman and Rett syndromes and is being evaluated for other disorders. The ORCA T-score ranges from 25.8 to 83.8, with higher ORCA T-scores indicate greater communication ability.
Neurodevelopmental Function as measured by the Vineland Adaptive Behavior Scales | Baseline to 24 months
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3), is a standardized, validated, and reliable assessment tool designed to measure the adaptive behavior of individuals from birth through adulthood through multiple domains, including communication and socialization. The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better adaptive functioning.
Neurodevelopmental Function as measured by the Bayley Scales of Infant and Toddler Development | Baseline to 24 months
  The Bayley Scales of Infant and Toddler Development is a standardized, validated, and reliable assessment tool for evaluating developmental functioning in infants and toddlers across subdomains of cognition and language (receptive and expressive communication). The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better neurodevelopment.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Kim-McManus, M.D., Principal Investigator — UCSD Rady Children's Hospital
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No